CLINICAL TRIAL: NCT06529380
Title: A Randomized Trial of Deep Brain Stimulation of the Nucleus Accumbens for Severe Self-Injurious Behaviours in Children
Brief Title: Deep Brain Stimulation for Severe Self-Injurious Behaviour in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, George Ibrahim, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REB # 1000081171
Record Dates: First submitted 2024-02-26; First posted 2024-07-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Self-Injurious Behavior; Autism Spectrum Disorder
Keywords: deep brain stimulation; DBS; ASD; SIB; nucleus accumbens
MeSH Terms: conditions — Self-Injurious Behavior; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (DBS ON, then OFF) (Active Comparator): Group 1: DBS will be switched ON in Block 1 (three months) after the initial four-week post-operative period. The DBS device will then be turned OFF for two weeks ("washout period"). The device will remain OFF in Block 2 (three months).
  Interventions: Device: DBS ON; Device: DBS OFF
- Group 2 (DBS OFF, then ON) (Placebo Comparator): Group 2: DBS will remain OFF in Block 1 (three months) after the initial four-week post-operative period. The device will remain off for two weeks thereafter ("washout period"). DBS will be switched ON in Block 2 (three months).
  Interventions: Device: DBS ON; Device: DBS OFF

INTERVENTIONS:
Device: DBS ON — Electrical stimulation of the nucleus accumbens.
Device: DBS OFF — DBS will remain OFF (on at 0V).

SUMMARY:
Deep Brain Stimulation for the Treatment of Severe Refractory Self-Injurious Behaviour in Children with Autism Spectrum Disorder: A Randomized Trial

To evaluate the effectiveness of deep brain stimulation (DBS) of the nucleus accumbens for the treatment of severe refractory, repetitive self-injurious behavior (SIB) in children with Autism Spectrum Disorder. Secondary objectives are to examine the effects of DBS on subtypes of SIB through functional analysis.

DETAILED DESCRIPTION:
The proposed study is a single-center, double-blinded, block-randomized crossover trial.

Twenty-five (25) participants will be recruited and enrolled in this trial to undergo bilateral nucleus accumbens DBS. After recovery, participants will be randomized to a 3 month block of active stimulation or the DBS will remain off. After a two week washout period, the participants will cross over to the other group. At the end of the second block, all patients will have their DBS devices activated during an open label period. All participants will have baseline assessments that will be repeated at the end of each block.

Expected study duration is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-17 at the time of enrollment
* DSM-5 diagnosis of Autism Spectrum Disorder
* History of repetitive self-injurious behaviour, as reported by parents and documented on clinical assessment, either at the time of enrollment into the study or in prior medical records. The definition of self-injury is contextual, but requires ongoing, intermittent or continuous manifestation of self-mediated physical injury to the child.
* Foreseeable risk of serious future self-harm.
* Screening by study team for presence automatically reinforced self-injurious behaviour (ASIB) subtype 2 or subtype 3 based on caregiver history.
* Failure or non-eligibility of medical therapy with ongoing repetitive self-injurious behaviours, at 6 months or more after initiation of therapy.
* Parents or legal guardians, including caregivers, informed and able to provide written consent.
* Able to comply with all testing, follow-up visits, and study appointments and protocols for 12 months following the end of the duration of the study.

Exclusion Criteria:

* Substance dependence or abuse in the last 6 months, excluding caffeine and nicotine.
* Any contraindication to MRI scanning.
* Presence of cardiac arrhythmias, or other cardiac, respiratory, renal or endocrine conditions that may incur significant risk from a surgical procedure.
* Pregnancy.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Repetitive Behaviors Scale-Revised (RBS-R) | Baseline, 4 weeks, 16 weeks, 30 weeks, 52 weeks
  A 44-item questionnaire that asks parents/caregivers how often a particular behaviour is seen occurring in the participant on a scale of 0-3, as well as a summary measure of how often the repetitive behaviours occur overall on a scale of 1-100.
  Higher scores indicate greater severity.

SECONDARY OUTCOMES:
Self-injurious behaviour log | Baseline (3 months), weekly during trial
  Parent/caregiver-reported frequency of repetitive self-injurious events over a given time period (i.e. number of events per day)
Repetitive Behaviour Questionnaire-2 (RBQ-2) | Baseline, 4 weeks, 16 weeks, 30 weeks, 52 weeks
  A 20-item parent/caregiver questionnaire that measures the frequency of a child's repetitive, restricted, and sensory behaviours.
  Questionnaire scores can be added to give a Total Repetitive Behaviours Score, within a minimum score of 20 and a maximum score of 60 (with responses '3' and '4' combined).
  Higher scores indicate greater severity.
Self-Injurious Behavior Questionnaire (SIB-Q) | Baseline, 4 weeks, 16 weeks, 30 weeks, 52 weeks
  A 25-item scale with Likert-style response options that measures self-injurious behavior among those with developmental disabilities.
  Scores range from 0 to 100, with higher scores indicating greater severity.
Pediatric Quality of Life Inventory (PedsQL) Questionnaire | Baseline, 4 weeks, 16 weeks, 30 weeks, 52 weeks
  A parent questionnaire designed to evaluate health-related quality of life in children.
  Scores range from 0 to 92, with higher scores indicating poorer quality of life.
Autism Diagnostic Observation Schedule (ADOS) Assessment questionnaire | Baseline, 16 weeks, 30 weeks
  A standardized, activity-based assessment designed to evaluate communication skills, social interaction, and imaginative use of materials in individuals who are suspected to have autism spectrum disorder.
  Classifications:
  * Non-spectrum: communication <1, social interaction <3, communication + social <6
  * Autism spectrum: communication >2, AND social interaction >4, AND communication + social 7-9
  * Autism: communication >3, AND social interaction >6, AND communication + social >10
  Higher scores indicate a greater presence of behaviours associated with autism spectrum disorder.
Modified Overt Aggression Scale (MOAS) questionnaire | Baseline, 4 weeks, 16 weeks, 30 weeks, 52 weeks
  A brief survey of overt aggression. Scores range from 0 to 40, with higher scores indicating greater severity.
The Burden Scale for Family Caregivers - Short Version (BSFC-S) questionnaire | Baseline, 4 weeks, 16 weeks, 30 weeks, 52 weeks
  A brief survey of parental burden of care. Scores range from 0 to 30, with higher scores indicating a greater burden.
Functional analysis (FA) assessment | Baseline, 16 weeks, 30 weeks
  An observation-based behavioural assessment that requires observing and quantifying how self-injurious behaviour (SIB) changes across conditions of a standardized and replicable assessment.

CONTACTS AND LOCATIONS:
Overall Officials: George M Ibrahim, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada